CLINICAL TRIAL: NCT06196853
Title: Nephroprotective Effects of Aminophylline in Pediatric Oncologic Patient on Cisplatin Based Chemotherapy; Double Blind Randomized Controlled Trial
Brief Title: Prevention of Cisplatin-induced Nephrotoxicity
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4639141
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury; Renal Tubulopathy
Keywords: Acute Kidney Injury; Chemotherapy induced kidney related complication
MeSH Terms: conditions — Acute Kidney Injury | interventions — Aminophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): 5%DNSS/2 with KCL and MgSO4 IV infusion with rate 125 ml/m2/hr.
- Treatment (Experimental): 5%DNSS/2 with KCL and MgSO4 IV infusion with rate 125 ml/m2/hr. plus aminophylline.
  Interventions: Drug: Aminophylline

INTERVENTIONS:
Drug: Aminophylline — Give aminophylline for 5 days to keep serum theophylline level 5-15 mg/dl
  Arms: Treatment

SUMMARY:
The research design is a prospective, randomized, controlled clinical trial in children to study effect of aminophylline in preserving renal function in oncologic patient received cisplatin either combined with other CMT or used alone. The participants in both groups will receive standard protocol pre-cisplatin infusion which include hydration with 5%DNSS/2 with KCL and MgSO4 IV infusion. In the treatment group, the participants will receive aminophylline infusion in the first 24 hours along with cisplatin, followed by oral aminophylline oral three times daily orally for 4 consecutive days post cisplatin. The aminophylline serum level will be maintained at the therapeutic range 10-20 mg. The side effect of aminophylline including nausea, vomiting and ECG will be monitored. The collected data including urine volume, GFR (estimated by cystatin C-creatinine based equation and by radiopharmaceutical-Tc DTPA), and renal tubular biomarker (urine B2 macroglobulin and urine NGAL) will be collected at baseline before receiving cisplatin, 24 hours and 5 days post cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18 years old
* Oncology patients who receive cisplatin-based therapy

Exclusion Criteria:

* Preexisting renal anomalies
* Preexisting GFR less than 60 ml/min/1.73 m2
* Contraindication of aminophylline including structural heart disease, arrhythmia, hyperthyroidism, chronic liver disease, epilepsy
* Aminophylline use within 24 hours prior to study entry

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in glomerular filtration rate | Baseline before cisplatin, and 48 hours 72 hours and 21 days post cisplatin
  Glomerular filtration rate is calculated using Cystatin C-creatinine-based equations. (ref. Kidney Int. 2012 Aug;82(4):445-53.)

SECONDARY OUTCOMES:
Renal tubular biomarkers | Baseline before cisplatin, and 48 hours 72 hours and 21 days post cisplatin
  Urine for beta2 macroglobulin

CONTACTS AND LOCATIONS:
Overall Officials: Anirut Pattaragarn, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Mahidol university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McSweeney KR, Gadanec LK, Qaradakhi T, Ali BA, Zulli A, Apostolopoulos V. Mechanisms of Cisplatin-Induced Acute Kidney Injury: Pathological Mechanisms, Pharmacological Interventions, and Genetic Mitigations. Cancers (Basel). 2021 Mar 29;13(7):1572. doi: 10.3390/cancers13071572. PMID 33805488
- [Background] Sugawara M, Mochizuki T, Takekuma Y, Miyazaki K. Structure-affinity relationship in the interactions of human organic anion transporter 1 with caffeine, theophylline, theobromine and their metabolites. Biochim Biophys Acta. 2005 Aug 15;1714(2):85-92. doi: 10.1016/j.bbamem.2005.06.006. PMID 16038872
- [Background] Alsaadoun S, Rustom F, Hassan HA, Alkhurais H, Aloufi M, Alzahrani S, Bakhsh S, Dalbhi SA. Aminophylline for improving acute kidney injury in pediatric patients: A systematic review and meta-analysis. Int J Health Sci (Qassim). 2020 Nov-Dec;14(6):44-51. PMID 33192231
- [Background] Benoehr P, Krueth P, Bokemeyer C, Grenz A, Osswald H, Hartmann JT. Nephroprotection by theophylline in patients with cisplatin chemotherapy: a randomized, single-blinded, placebo-controlled trial. J Am Soc Nephrol. 2005 Feb;16(2):452-8. doi: 10.1681/ASN.2004030225. Epub 2004 Dec 8. PMID 15590762